CLINICAL TRIAL: NCT06923475
Title: Neoadjuvant Gemcitabine and Cisplatin in Combination With Perioperative Pembrolizumab Versus Upfront Surgery for Patients With Primary Resectable and Borderline Resectable Perihilar and Distal Cholangiocarcinoma (NEODISCO): A Multicentre Phase 2B/3 Randomized Controlled Trial
Brief Title: Neoadjuvant Gemcitabine and Cisplatin in Combination With Perioperative Pembrolizumab Versus Upfront Surgery for Patients With Primary Resectable and Borderline Resectable Perihilar and Distal Cholangiocarcinoma
Acronym: NEODISCO
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Maastricht University Medical Center (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Trial Office Medical Oncology VUmc, Prof. Dr. J.W. Wilmink, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-516898-72-00; R-000724 (Other Grant/Funding Number: Merck Sharp & Dohme)
Record Dates: First submitted 2025-02-25; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-02

CONDITIONS: Extrahepatic Cholangiocarcinoma; Perihilar Cholangiocarcinoma; Distal Cholangiocarcinoma; Resectable; Borderline Resectable
Keywords: Extrahepatic cholangiocarcinoma; Perihilar Cholangiocarcinoma; Distal Cholangiocarcinoma; Resectable; Borderline resectable
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Neoadjuvant gemcitabine plus cisplatin in combination with perioperative pembrolizumab (Intervention)
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine, Cisplatin
- Arm B (No Intervention): Upfront surgery (Standard of care)

INTERVENTIONS:
Drug: Pembrolizumab — Patients will initiate with 2 sets of 3 cycles of neoadjuvant gemcitabine and cisplatin in combination with perioperative pembrolizumab (up to total of 1 year immunotherapy treatment)
  Arms: Arm A
Drug: Gemcitabine, Cisplatin — Patients will initiate with 2 sets of 3 cycles of neoadjuvant gemcitabine and cisplatin in combination with perioperative pembrolizumab (up to total of 1 year immunotherapy treatment)
  Arms: Arm A

SUMMARY:
Extrahepatic cholangiocarcinoma (eCCA) is a rare and aggressive cancer with poor prognosis. ECCA can be further subcategorised in perihilar and distal cholangiocarcinoma (pCCA and dCCA). Surgical resection is the only potential cure, but only one-third of patients are eligible. Even among those deemed resectable, a significant portion (≈30%) experience disease progression before surgery, while another 30% are found unresectable during exploration. High recurrence rates and postoperative complications further limit survival, with 5-year overall survival ranging from 13% (R1 resection) to 40% (R0 resection). Given the long preoperative work-up period and lack of treatment during this phase, a neoadjuvant approach may improve outcomes by increasing R0 resections, reducing recurrence, and optimizing patient selection.

This multicenter, randomized phase 2B/3 trial aims to assess whether neoadjuvant gemcitabine and cisplatin plus perioperative pembrolizumab improves event-free survival in patients with resectable and borderline resectable pCCA and dCCA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed resectable or borderline resectable pCCA and dCCA. These are all the patients considered candidates for upfront surgical exploration, with intent to resect, as confirmed by local MDT and the study expert panel also taking into consideration endoscopic and radiological findings. In cases where drainage is not required, patients with a disease highly suspicious for extrahepatic cholangiocarcinoma, as determined by the expert MDT, may be included without histological proof to prevent unnecessary post-ERCP complications.
* Successful drainage, in case of clinical significant bile duct obstruction.
* MidCCA inclusion in the NEODISCO-trial will be permitted and will be included according to the proposed type of resection.
* Male/female participants who are at least 18 years of age on the day of signing informed consent.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.

Exclusion Criteria:

* Upfront "clearly" unresectable pCCA: circumferential unreconstructable vascular involvement of the FLR and/or insufficient FLR for potential radical resection. Insufficient FLR is defined as <30% residual volume or a function <2.7 min/m2. Patients considered borderline resectable but, by the discretion of the MDT, not a candidate for upfront exploration/resection, are considered ineligible for NEODISCO.
* Upfront clearly unresectable dCCA (following DPCG criteria).
* Patients with proven N2 lymph nodes (according to the AJCC 8th edition).
* PCCA eligible for liver transplantation.
* Intrahepatic cholangiocarcinoma with hilar involvement.
* Cancer suspicious for ampullary carcinoma (for instance involvement of papilla during endoscopy).
* Local recurrence following prior resection of eCCA (patients who develop local recurrence during the study are however not excluded).
* Patients with underlying liver diseases: PSC, untreated hepatitis, cirrhosis child-Pugh B, C.
* Previous malignancy unless no evidence of disease, or diagnosed more than 3 years before diagnosis of eCCA, or with a life expectancy of more than 5 years from date of inclusion.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2028-11-06 (Estimated); Study Completion 2028-11-06 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 18 months
  An event is defined as the time from randomization to any progression of disease leading to unresectability, progression or recurrence of disease after surgery (all based on RECIST or pathology) or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Median, 2-, 3-, 5- years OS
  Most important secondary endpoint: median OS defined as the time from randomization to death due to any cause. 2-, 3- and 5-years OS will also be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF